CLINICAL TRIAL: NCT00948766
Title: A 24 Week, Prospective, Randomized, Parallel-group, Double-blind, Multi-center Study (ENA713DUS44) Comparing the Effects of Rivastigmine Patch 15 cm^2 vs. Rivastigmine Patch 5 cm^2 on ACTivities of Daily Living and CognitION in Patients With Severe Dementia of the Alzheimer's Type (ACTION) and a 24-week Open-label Extension to Study ENA713DUS44
Brief Title: Effects of Rivastigmine Patch on Activities of Daily Living and Cognition in Patients With Severe Dementia of the Alzheimer's Type (ACTION) (Study Protocol CENA713DUS44, NCT00948766) and a 24 Week Open-label Extension to Study CENA713DUS44
Acronym: ACTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CENA713DUS44; NCT01054755 (obsolete NCT alias)
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; dementia; Alzheimer's type
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Rivastigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Rivastigmine 13.3 mg/24 h transdermal patch (Experimental): In the core study, patients were titrated to the rivastigmine 13.3 mg/24 h dose in 2 steps. For Weeks 1-4, patients received rivastigmine 4.6 mg/24 h. For Weeks 5-8, patients received rivastigmine 9.5 mg/24 h and placebo. For Weeks 9-24, patients received rivastigmine 13.3 mg/24 h and placebo. In the extension study, all patients were switched to rivastigmine 9.5 mg/24 h for a 4-week titration period and were then titrated up to 13.3 mg/24 h for a further 20 weeks of treatment.
  Interventions: Drug: Rivastigmine 4.6 mg/24 h (5 cm^2); Drug: Rivastigmine 9.5 mg/24 h (10 cm^2); Drug: Rivastigmine 13.3 mg/24 h (15 cm^2); Drug: Placebo
- Rivastigmine 4.6 mg/24 h transdermal patch (Active Comparator): In the core study, patients received rivastigmine 4.6 mg/24 h daily. For Weeks 1-4, patients received rivastigmine 4.6 mg/24 h. For Weeks 5-24, patients received rivastigmine 4.6 mg/24 h and placebo. No patients received this treatment in the extension study.
  Interventions: Drug: Rivastigmine 4.6 mg/24 h (5 cm^2); Drug: Placebo

INTERVENTIONS:
Drug: Rivastigmine 4.6 mg/24 h (5 cm^2) — Rivastigmine was supplied in a 5 cm^2 patch which released 4.6 mg/24 h. Patches were changed daily.
  Other Names: ENA713D; Exelon; Exelon patch
Drug: Rivastigmine 9.5 mg/24 h (10 cm^2) — Rivastigmine was supplied in a 10 cm^2 patch which released 9.5 mg/24 h. Patches were changed daily.
  Other Names: ENA713D; Exelon; Exelon path
  Arms: Rivastigmine 13.3 mg/24 h transdermal patch
Drug: Rivastigmine 13.3 mg/24 h (15 cm^2) — Rivastigmine was supplied in a 15 cm^2 patch which released 13.3 mg/24 h. Patches were changed daily.
  Other Names: ENA713D; Exelon; Exelon patch
  Arms: Rivastigmine 13.3 mg/24 h transdermal patch
Drug: Placebo — Placebo patches were identical in size and composition to the corresponding rivastigmine patches, except that they did not contain rivastigmine. Patches were changed daily.

SUMMARY:
The core study assessed the efficacy of a higher dose of rivastigmine 13.3 mg/24 h transdermally (15 cm^2 patch) compared to a lower dose of the rivastigmine 4.6 mg/24 h transdermally (5 cm^2 patch) in patients with Severe Dementia of the Alzheimer's Type in a 24-week study. The extension study obtained additional safety and efficacy data, as well as provided the higher dose rivastigmine patch to all patients who completed the core study for an additional 24 weeks.

ELIGIBILITY:
Core study

Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease (AD) according to National Institute of Neurological Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria.
* A Mini-Mental State Examination (MMSE) score of ≥ 3 and ≤ 12.
* Be able to complete at least 1 item on the Severe Impairment Battery (SIB).
* Residing with someone in the community or in regular contact with the primary caregiver.
* Be ambulatory or ambulatory with aid.

Exclusion Criteria:

* An advanced, severe, progressive, or unstable disease of any type that may interfere with efficacy and safety assessments or put the patient at special risk.
* Patients currently residing in a nursing home.
* Any current medical or neurological condition other than AD that could explain the patient's dementia.
* A current diagnosis of probable or possible vascular dementia.
* A current diagnosis of severe or unstable cardiovascular disease.
* A current diagnosis of bradycardia (< 50 beats per minute [bpm]), sick-sinus syndrome, or conduction defects.
* Clinically significant urinary obstruction.
* History of malignancy of any organ system within the past 5 years unless patient is verified to be in stable condition with no active metastasis.
* Current diagnosis of an active skin lesion/disorder that would prevent the patient from using a transdermal patch every day.
* A known exaggerated pharmacological sensitivity or hypersensitivity to drugs similar to rivastigmine, or to other cholinergic compounds.
* Taken any of the following substances (at the time of the Baseline Visit [Visit 2]).
* Succinylcholine-type muscle relaxants during the previous 2 weeks.
* Lithium during the previous 2 weeks.
* An investigational drug during the previous 4 weeks.
* A drug or treatment known to cause major organ system toxicity during the previous 4 weeks.
* Rivastigmine (oral or transdermal patch), donepezil, galantamine, other cholinesterase inhibitors (eg, tacrine, physostigmine, or pyridostigmine), or other approved treatments for Alzheimer's disease during the previous 2 weeks, with exception of stable treatment with memantine for at least 3 months before study entry (Visit 1).
* Centrally acting anticholinergic drugs including tricyclic and tetracyclic antidepressants during the previous 4 weeks.
* Selegiline unless taken at a stable dose during the previous 4 weeks.
* Peripheral anticholinergics not taken at a stable dose during the previous 4 weeks.

Extension study

Inclusion Criteria:

* Complete the double-blind phase (Week 24) of the core study.
* Provide, if mentally competent, a separate written informed consent prior to participation in the extension study. In addition, the patient's caregiver, will provide written informed consent prior to the patient's participation in the open-label extension study. If the patient is not able to provide written informed consent, written informed consent must be obtained from the legally authorized representative on the patient's behalf.
* Continue to reside with someone in the community or in regular contact with the primary caregiver; patients who reside in an assisted living facility are eligible to participate.
* Continue to have a primary caregiver willing to accept responsibility for supervising treatment (eg, application and removal of the patch daily at approximately the same time of day), assessing the condition of the patient throughout the extension study.
* Must be medically stable and tolerating the current dose of rivastigmine patch as determined by the investigator.

Exclusion Criteria:

Refer to the core study protocol for full details of the exclusion criteria.

* Patients who discontinued the core study due to any reason are excluded.
* No additional exclusions may be applied by the investigator, in order to ensure that the study population will be representative of all eligible patients.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Actual)
Dates: Start 2009-07; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (95):
- United States (93):
  - Clinical Research Advantage Inc./Neurological. Physicians of Arizona, Inc, Tempe, Arizona
  - Northwest Neuro Specialist, PLLC, Tucson, Arizona
  - IHS Research Center Inc., Conway, Arkansas
  - East Bay Physicians Medical Group, Berkeley, California
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Neuro Pain Medical Center, Fresno, California
  - Margolin Brain Institute, Fresno, California
  - Collaborative Neuroscience Network Inc., Garden Grove, California
  - PCND Neuroscience Research Institute Inc./The Center for Memory and Aging, Poway, California
  - Anderson Clinical Research, Redlands, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - California Neuroscience Research Medical Group, Inc., Sherman Oaks, California
  - Viking Clinical Research Center, Temecula, California
  - Collaborative Neuroscience Network, Inc, Torrance, California
  - Senior Care of Colorado, Aurora, Colorado
  - Clinical Research Studies Dept. of Clinical Science and Medical Education, Boca Raton, Florida
  - Quantum Laboratories Memory Disorder Center, Deerfield Beach, Florida
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Neurologic Consultants, PA, Fort Lauderdale, Florida
  - White-Wilson Medical Center, Fort Walton Beach, Florida
  - MD Clinical, Hallandale, Florida
  - Sunrise Clinical Research, Inc, Hollywood, Florida
  - Compass Research, LLC, Orlando, Florida
  - Integrity Research, LLC, Pensacola, Florida
  - Neurostudies, Inc., Port Charlotte, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - Center for Clinical Trials, Venice, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Alexian Brothers Neuroscience Institute, Elk Grove Village, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - MidAmerica Neuroscience Reseach Institute, Lenexa, Kansas
  - Precise Clinical Research Solutions, Manhattan, Kansas
  - LSU Health Sciences Center/Department of Psychiatry Psychopharmacology Research Clinic, Shreveport, Louisiana
  - J. Gary Booker, MD APMC, Shreveport, Louisiana
  - Pharmasite Research, Baltimore, Maryland
  - The Samuel and Alexia Bratton Memory Clinic, William Hill Inc, Easton, Maryland
  - Neuroscience Research of the Berkshires, Pittsfield, Massachusetts
  - Michigan Neurology Associates, P.C., Clinton Township, Michigan
  - Wayne State University/Detroit Medical center, Detroit, Michigan
  - West Michigan Clinical Research, Muskegon, Michigan
  - Orr & Associates Memory and Geriatric Behavioral Health Clinic, Saint Paul, Minnesota
  - Neurological Research Clinic, Hattiesburg Clinic, Hattiesburg, Mississippi
  - The Neuroscience Center, Ocean Springs, Mississippi
  - St. Louis University, St Louis, Missouri
  - Sky, LLC., St Louis, Missouri
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - NeuroCognitive Institute, Mount Arlington, New Jersey
  - UMDNJ-Robert Wood Johnson Medical Center, New Brunswick, New Jersey
  - Alzheimer's Research Corporation, Paterson, New Jersey
  - UMDNJ-School of Osteopathic Medicine Center, Stratford, New Jersey
  - Memory Enhancement Center of NJ, Toms River, New Jersey
  - Upstate Clinical Research, LLC, Albany, New York
  - Dent Neurological Institute, Amherst, New York
  - Neurological Care of Central NY, Liverpool, New York
  - Eastside Comprehensive medical Center, LLC, New York, New York
  - Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York
  - Behavioral Medical Research of Staten Island, Staten Island, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - The Burke Rehabilitation Hospital, White Plains, New York
  - Alzheimer's Memory Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Clinical Trials of America, Inc., Winston-Salem, North Carolina
  - Valley Medical Research, Centerville, Ohio
  - University Neurology, Inc., Cincinnati, Ohio
  - Cognitive Assessment Clinic, Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Paramount Clinical Research, Bridgeville, Pennsylvania
  - Department of Veterans Affairs Medical Center, Coatesville, Pennsylvania
  - Westmoreland Neurology associates, Inc., Greensburg, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Research Protocol Management Specialists, Pittsburgh, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Psychiatric Consultants, PC, Franklin, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Jacinto Medical Group, PA, Baytown, Texas
  - Future Search Trials, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Radiant Research Inc., San Antonio, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - The Memory Clinic, Bennington, Vermont
  - TLC Neurology, P.L.L.C, Arlington, Virginia
  - UVA Neurology, Charlottesville, Virginia
  - Neurological Associates, Inc., Richmond, Virginia
  - Alliance Research Group, LLC, Richmond, Virginia
  - The Center for Excellence in Aging and Geriatric Health, Williamsburg, Virginia
  - Internal Medicine Northwest, Tacoma, Washington
  - Independent Psychiatric Consultants, SC, Waukesha, Wisconsin
- Puerto Rico (2):
  - Metro Medical Center, Bayamón
  - INSPIRA Clinical Research, San Juan

REFERENCES:
- [Derived] Grossberg GT, Farlow MR, Meng X, Velting DM. Evaluating high-dose rivastigmine patch in severe Alzheimer's disease: analyses with concomitant memantine usage as a factor. Curr Alzheimer Res. 2015;12(1):53-60. doi: 10.2174/1567205011666141218122835. PMID 25523430

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient in each treatment group in the core study and one patient in the treatment group in the extension study did not receive study medication; they were not included in the safety set.
Groups:
- Rivastigmine 13.3 mg/24 h Transdermal Patch: Patients received rivastigmine 13.3 mg/24 h (15 cm^2).
- Rivastigmine 4.6 mg/24 h Transdermal Patch: Patients received rivastigmine 4.6 mg/24 h (5 cm^2).
Period: Core Study
Arm/Group | Rivastigmine 13.3 mg/24 h Transdermal Patch | Rivastigmine 4.6 mg/24 h Transdermal Patch
Started | 356 | 360
Exposed to Study Medication | 355 | 359
Completed | 229 | 234
Not Completed | 127 | 126
Not completed — Adverse Event | 73 | 51
Not completed — Unsatisfactory Therapeutic Effect | 13 | 14
Not completed — Patient Withdrew Consent | 27 | 46
Not completed — Lost to Follow-up | 3 | 2
Not completed — Administrative Problems | 2 | 2
Not completed — Death | 1 | 1
Not completed — Protocol Deviation | 8 | 10
Period: Extension Study
Arm/Group | Rivastigmine 13.3 mg/24 h Transdermal Patch | Rivastigmine 4.6 mg/24 h Transdermal Patch
Started | 397 (397 of the 463 patients who completed the core study entered the extension study.) | 0 (No patients received this treatment in the extension study.)
Exposed to Study Medication | 396 | 0
Completed | 306 | 0
Not Completed | 91 | 0
Not completed — Adverse Event | 43 | 0
Not completed — Unsatisfactory Therapeutic Effect | 2 | 0
Not completed — Study Drug No Longer Required | 1 | 0
Not completed — Patient Withdrew Consent | 32 | 0
Not completed — Lost to Follow-up | 8 | 0
Not completed — Administrative Problems | 1 | 0
Not completed — Death | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Core Study: Rivastigmine 13.3 mg/24 h Transdermal Patch: Patients received rivastigmine 13.3 mg/24 h (15 cm^2).
- Core Study: Rivastigmine 4.6 mg/24 h Transdermal Patch: Patients received rivastigmine 4.6 mg/24 h (5 cm^2).
- Total: Total of all reporting groups
Arm/Group | Core Study: Rivastigmine 13.3 mg/24 h Transdermal Patch | Core Study: Rivastigmine 4.6 mg/24 h Transdermal Patch | Total
Number analyzed (Participants) | 356 | 360 | 716
Age Continuous [Mean (Standard Deviation); unit: years] | 77.6 (8.69) | 76.5 (9.35) | 77.0 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 227 | 234 | 461
  Male | 129 | 126 | 255

OUTCOME MEASURES:

1. Primary Outcome: Core Study: Change From Baseline in the Alzheimer's Disease Cooperative Study-Activities of Daily Living-Severe Impairment Version (ADCS-ADL-SIV) Score at Week 24
Description: The ADCS-ADL-SIV is designed to assess the patient's performance of both basic and instrumental activities of daily living such as those necessary for personal care, communicating and interacting with other people, maintaining a household, conducting hobbies and interests, and making judgments and decisions. For each of the 19 questions in the ADCS-ADL-SIV, there was either a forced choice of best response or a "yes" or "no" question with additional sub-questions. Responses for each item were obtained from the caregiver through an interview. Higher numbered scores and answers of "yes" reflected a more self-sufficient individual. The total score was calculated as the sum of all items and sub-questions and ranged from 0 to 54. A higher total score represented a higher functioning patient. A positive change score indicates improvement.
Time Frame: Baseline of the core study to Week 24 of the core study
Population: Modified full analysis set: All randomized patients who received at least 1 dose of study medication and had at least 1 post-baseline measurement of the co-primary efficacy variables. Only patients with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rivastigmine 13.3 mg/24 h Transdermal Patch | Rivastigmine 4.6 mg/24 h Transdermal Patch
Number analyzed (Participants) | 310 | 303
Units on a scale | -2.6 (6.82) | -3.6 (7.68)

2. Primary Outcome: Core Study: Change From Baseline in the Severity Impairment Battery (SIB) Score at Week 24
Description: The SIB is a 40-item scale developed for the evaluation of the severity of cognitive dysfunction in more advanced Alzheimer Disease patients. The domains assessed included social interaction, memory, language, attention, orientation, praxis, visuo-spatial ability, construction, and orienting to name. The items of the SIB were developed as simple 1-step commands which are presented by a trained rater with gestural cues and repeated if necessary. The SIB was scored from 0 to 100, with higher scores reflecting higher levels of cognitive ability. A positive change score indicates improvement.
Time Frame: Baseline of the core study to Week 24 of the core study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rivastigmine 13.3 mg/24 h Transdermal Patch | Rivastigmine 4.6 mg/24 h Transdermal Patch
Number analyzed (Participants) | 313 | 316
Units on a scale | -1.6 (13.54) | -6.4 (14.01)

3. Secondary Outcome: Core Study: Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) Score at Week 24
Description: The ADCS-CGIC assesses the clinical meaningfulness of a treatment based on the clinician's rating of change. The rating is provided by a trained clinician or psychometrician blinded to the patient's treatment. The rater interviewed the patient and caregiver separately at Baseline using a worksheet that provided space for notes and comments. At baseline, raters had access to all of the patient's available records and evaluations. The rater used a similar worksheet at follow-up visits, and referred to the baseline worksheet prior to making a rating of change. The worksheets were divided into 3 domains: mental/cognitive state, behavior, and functioning. Change ratings were based on a 7-point scale: Marked (1), moderate (2), and minimal improvement (3), no change (4), and marked (5), moderate (6), and minimal worsening (7). The percentage of patients in each of the 7 categories is reported.
Time Frame: Baseline of the core study to Week 24 of the core study
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Rivastigmine 13.3 mg/24 h Transdermal Patch | Rivastigmine 4.6 mg/24 h Transdermal Patch
Number analyzed (Participants) | 313 | 315
Percentage of patients
  Marked improvement | 1.0 | 1.3
  Moderate improvement | 3.5 | 3.5
  Minimal improvement | 20.1 | 11.4
  No change | 34.2 | 29.2
  Minimal worsening | 24.3 | 31.4
  Moderate worsening | 14.1 | 19.0
  Marked worsening | 2.9 | 4.1

4. Secondary Outcome: Core Study: Change From Baseline in the Neuropsychiatric Inventory (NPI-12) Score at Week 24
Description: The NPI-12 assesses a wide range of behaviors encountered in patients with dementia to provide a means of distinguishing the frequency and severity of behavioral changes over time. Ten behavioral and 2 neurovegetative domains were evaluated in an interview with the caregiver given by a mental health professional. The scale included both frequency and severity ratings of each domain as well as a composite domain score (frequency x severity). The sum of the composite scores for the 12 domains yielded the NPI-12 total score. The NPI-12 was scored from 0 to 144, with lower scores reflecting improvement in psychiatric behavior. A negative change score indicates improvement.
Time Frame: Baseline of the core study to Week 24 of the core study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rivastigmine 13.3 mg/24 h Transdermal Patch | Rivastigmine 4.6 mg/24 h Transdermal Patch
Number analyzed (Participants) | 313 | 313
Units on a scale | -0.4 (14.01) | 1.2 (16.79)

5. Secondary Outcome: Extension Study: Change From Baseline in the Alzheimer's Disease Cooperative Study-Activities of Daily Living-Severe Impairment Version (ADCS-ADL-SIV) Score at Week 24
Description: as for outcome 1
Time Frame: Baseline of the core study to Week 24 of the extension study
Population: Modified full analysis set: All patients who received at least 1 application of study medication and had at least 1 efficacy assessment in the extension study. Only patients with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rivastigmine 13.3 mg/24 h Transdermal Patch
Number analyzed (Participants) | 372
Units on a scale | -4.3 (8.37)

6. Secondary Outcome: Extension Study: Change From Baseline in the Severity Impairment Battery (SIB) Score at Week 24
Description: as for outcome 2
Time Frame: Baseline of the core study to Week 24 of the extension study
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rivastigmine 13.3 mg/24 h Transdermal Patch
Number analyzed (Participants) | 379
Units on a scale | -5.9 (16.72)

7. Secondary Outcome: Extension Study: Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) Score at Week 24
Description: as for outcome 3
Time Frame: Baseline of the core study to Week 24 of the extension study
Population: as for outcome 5
Measure: Number; unit: Percentage of patients
Arm/Group | Rivastigmine 13.3 mg/24 h Transdermal Patch
Number analyzed (Participants) | 381
Percentage of patients
  Marked improvement | 1.8
  Moderate improvement | 5.0
  Minimal improvement | 9.7
  No change | 26.2
  Minimal worsening | 31.5
  Moderate worsening | 21.5
  Marked worsening | 4.2

ADVERSE EVENTS:
Time Frame: Adverse events were reported from randomization in the core study through the end of the extension study (48 weeks).
Description: Safety set: All patients who received at least 1 dose of study medication and had at least 1 safety assessment after baseline. One patient in each treatment group did not receive study medication and were not included in the safety set.
Groups:
- Extension Study: Rivastigmine 13.3 mg/24 h Transdermal Patch: Patients received rivastigmine 13.3 mg/24 h (15 cm^2).
Arm/Group | Core Study: Rivastigmine 13.3 mg/24 h Transdermal Patch | Core Study: Rivastigmine 4.6 mg/24 h Transdermal Patch | Extension Study: Rivastigmine 13.3 mg/24 h Transdermal Patch
Serious Adverse Events (participants affected / at risk) | 82/355 | 74/359 | 79/396
Other Adverse Events (participants affected / at risk) | 216/355 | 210/359 | 248/396
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Study: Rivastigmine 13.3 mg/24 h Transdermal Patch (N=355) | Core Study: Rivastigmine 4.6 mg/24 h Transdermal Patch (N=359) | Extension Study: Rivastigmine 13.3 mg/24 h Transdermal Patch (N=396)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 2
Bradycardia (Cardiac disorders) | 3 | 1 | 2
Bundle branch block left (Cardiac disorders) | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 3 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 1 | 2
Asthenia (General disorders) | 2 | 2 | 2
Chest discomfort (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 2 | 4 | 5
Fatigue (General disorders) | 0 | 1 | 1
Gait disturbance (General disorders) | 0 | 2 | 0
Malaise (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 2 | 3
Cellulitis (Infections and infestations) | 0 | 2 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Intestinal gangrene (Infections and infestations) | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 4 | 5 | 5
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 2 | 1 | 1
Urinary tract infection (Infections and infestations) | 5 | 7 | 8
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chemical poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 7 | 7 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 4 | 1 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 | 1 | 2
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 4 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 4 | 3 | 4
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 1
Blood pressure systolic decreased (Investigations) | 0 | 1 | 1
Cardiac enzymes increased (Investigations) | 1 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 6 | 4 | 6
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 4 | 1 | 4
Convulsion (Nervous system disorders) | 1 | 3 | 2
Coordination abnormal (Nervous system disorders) | 1 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 3 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 1
Dysstasia (Nervous system disorders) | 0 | 1 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Hypokinesia (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 2 | 2
Pneumocephalus (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 3 | 1
Somnolence (Nervous system disorders) | 0 | 2 | 2
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 7 | 6 | 7
Transient ischaemic attack (Nervous system disorders) | 4 | 1 | 4
Unresponsive to stimuli (Nervous system disorders) | 1 | 1 | 2
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 3 | 0
Agitation (Psychiatric disorders) | 2 | 6 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 3 | 1 | 2
Delirium (Psychiatric disorders) | 1 | 1 | 1
Depression (Psychiatric disorders) | 0 | 2 | 1
Major depression (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 3 | 6 | 5
Mutism (Psychiatric disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 | 1 | 0
Stress (Psychiatric disorders) | 1 | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 1 | 1
Rectocele (Reproductive system and breast disorders) | 1 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cystopexy (Surgical and medical procedures) | 1 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 1 | 1
Hysterectomy (Surgical and medical procedures) | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 2 | 0 | 1
Bloody discharge (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Haematoma (Vascular disorders) | 1 | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 1 | 3
Hypotension (Vascular disorders) | 0 | 3 | 2
Orthostatic hypotension (Vascular disorders) | 2 | 1 | 2
Shock (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core Study: Rivastigmine 13.3 mg/24 h Transdermal Patch (N=355) | Core Study: Rivastigmine 4.6 mg/24 h Transdermal Patch (N=359) | Extension Study: Rivastigmine 13.3 mg/24 h Transdermal Patch (N=396)
Diarrhoea (Gastrointestinal disorders) | 25 | 27 | 36
Nausea (Gastrointestinal disorders) | 23 | 17 | 19
Vomiting (Gastrointestinal disorders) | 27 | 24 | 30
Application site dermatitis (General disorders) | 30 | 36 | 43
Application site erythema (General disorders) | 48 | 44 | 52
Urinary tract infection (Infections and infestations) | 42 | 43 | 58
Fall (Injury, poisoning and procedural complications) | 30 | 26 | 42
Weight decreased (Investigations) | 37 | 26 | 47
Agitation (Psychiatric disorders) | 47 | 55 | 58
Anxiety (Psychiatric disorders) | 18 | 19 | 19
Depression (Psychiatric disorders) | 19 | 16 | 18
Hallucination (Psychiatric disorders) | 9 | 19 | 16
Insomnia (Psychiatric disorders) | 27 | 24 | 30
Urinary incontinence (Renal and urinary disorders) | 13 | 14 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.